CLINICAL TRIAL: NCT03428204
Title: Effect of Different Inflation Times on the Angiographic Result After Balloon Angioplasty in the Femoropopliteal Segment: a Prospective Randomized Clinical Trial
Brief Title: Effect of Inflation on the Angiographic Result After Balloon Angioplasty in the Femoropopliteal Segment
Acronym: Balloon-angio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/17AOU/406
Record Dates: First submitted 2017-12-08; First posted 2018-02-09 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Femoropopliteal Arterial Stenosis

STUDY DESIGN:
Intervention Model Description: The effect of two balloon inflation times will be evaluated in peripheral balloon angioplasty
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 180 seconds balloon dilation (Other): Percutaneous angioplasty with balloon dilation during 180 seconds for percutaneous treatment of femoropopliteal artery stenosis
  Interventions: Procedure: Balloon dilation during 180 seconds
- 300 seconds balloon dilation (Other): Percutaneous angioplasty with balloon dilation during 300 seconds for percutaneous treatment of femoropopliteal artery stenosis
  Interventions: Procedure: Balloon dilation during 300 seconds

INTERVENTIONS:
Procedure: Balloon dilation during 180 seconds — Percutaneous angioplasty with balloon dilation during 180 seconds as a method for percutaneous treatment of femoropopliteal artery lesions
  Other Names: Balloon dilation of femoropopliteal artery lesions during 180 seconds
  Arms: 180 seconds balloon dilation
Procedure: Balloon dilation during 300 seconds — Percutaneous angioplasty with balloon dilation during 300 seconds as a method for percutaneous treatment of femoropopliteal artery lesions
  Other Names: Balloon dilation of femoropopliteal artery lesions during 300 seconds
  Arms: 300 seconds balloon dilation

SUMMARY:
Percutaneous angioplasty with balloon dilation is the method of choice for the treatment of most femoropopliteal artery lesions. After balloon dilatation, arterial wall dissection with flow limiting dissection or recoil with residual stenosis often require additional procedures such as stent placement or prolonged balloon dilation. A shorter balloon inflation time of 30 sec will be accompanied by a higher number of flow limiting dissection or recoil, demanding a time consuming and expensive stent placement or balloon redilatation. The effect of different balloon inflation times has only been assessed ones in peripheral balloon angioplasty with better outcomes after prolonged balloon inflation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic atherosclerotic stenotic lesions of the femoropopliteal artery suitable for angioplasty in the adult population

Exclusion Criteria:

* Artery lesions shorter than 1 cm and longer than 10 cm length, total occlusions, severe calcification, previous angioplasty with current restenosis, previous stenting with current insistent restenosis and subintimal recanalization of the lesion
* No pregnant and nursing women will be included.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of residual stenosis between both groups | at 3 or 5 minutes
  The primary outcome of the study is to assess the difference in number of residual stenosis after balloon dilatation of the arterial lesion between both groups (3min and 5min). A residual stenosis (measured on the angiogram) responsible for an arterial stenosis of >30% will be defined as unsuccessful treatment.
  The group with the lowest number of arterial restenosis >30% after dilatation has the best primary outcome.

SECONDARY OUTCOMES:
Number of redilatation or additional stenting between both groups | at 3 or 5 minutes
  The secondary outcome of the study is to evaluate the difference in need of redilatation or provisional stenting after the first dilatation between both groups (3 vs 5min). If an arterial stenosis of >30% after dilatation is measured, a redilatation of an additional stenting will be placed. The group with the lowest number of redilatation or additional stenting after dilatation has the best secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Parla Astarci, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium